CLINICAL TRIAL: NCT04205188
Title: Do Therapeutic Exercises Improve Kinesiophobia and Health-Related Quality of Life in Adult Haemophilia Patients? A Randomized Controlled Trial.
Brief Title: The Effects of Therapeutic Exercises on Kinesiophobia in Haemophilic Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Volkan Deniz, PT (Other)
Responsible Party: Sponsor-Investigator, Volkan Deniz, PT, Director, Clinical Research, Cukurova University
Organization: Cukurova University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 89/56
Record Dates: First submitted 2019-12-13; First posted 2019-12-19 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Haemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercises and verbal information (Experimental): therapeutic exercises 3 days in a week and total 8 weeks and 60 minutes verbal information
  Interventions: Other: therapeutic exercises
- verbal information (No Intervention): 60 minutes information about effects of exercises on joint functions

INTERVENTIONS:
Other: therapeutic exercises — aerobic- balance -stretching and strengthening exercises
  Arms: exercises and verbal information

SUMMARY:
this study evaluates the effects of therapeutic exercises on kinesiophobia and health-related quality of life in adult haemophilia patients. half of participants will receive therapeutic exercises and verbal information about the positive effects of therapeutic exercises on physical pathologies due to hemophilic arthropathy while the other half will receive only verbal information.

DETAILED DESCRIPTION:
in haemophilia patients recurrent musculoskeletal hemorrhage cause to arthropathy characterized by severe degeneration of joint cartilage and bones. arthropathy leads to decrease in the patient's health related quality of life. furthermore pain, risk of injury and lack of motivation lead to decreased physical activity and development of kinesiophobia.

ELIGIBILITY:
Inclusion Criteria:

* Individuals older than 18 years
* diagnosed with hemophilia A or B
* having at least one joint with hemophilic arthropathy
* without cognitive problems
* speaking turkish

Exclusion Criteria:

* Individuals with another congenital coagulopathy such as Von Willebrand Syndrome,
* unable to walk due to hemophilic arthropathy
* developing inhibition against factor VIII-IX

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
tampa kinesiophobia scale | baseline, 8 weeks: change from baseline kinesiophobia at 8 weeks, 6 months: change from baseline kinesiophobia at 6 months
  This is a questionnaire consisting of a total of 17 questions evaluating fears related to pain or previous injury. participants can receive a maximum of 68 and minimum of 17 points in this questionnaire. there is a negative correlation between the score and kinesiophobia.
haemophilia adult health-related quality of life scale | baseline, 8 weeks: change from baseline health-related quality of life at 8 weeks, 6 months: change from baseline health-related quality of life at 6 months
  this questionnaire evaluates health-related quality of life in adult haemophilic individuals and consisting of ten sections -46 questions. participants can receive a maximum of 100 and a minimum of 0 points in this questionnaire. there is a negative correlation between the score and quality of life.

SECONDARY OUTCOMES:
short form-36 | baseline, 8 weeks: change from baseline health-related quality of life at 8 weeks, 6 months: change from baseline health-related quality of life at 6 months
  short form-36 is a quality of life questionnaire consisting of 8 sections and 36 questions. participants can receive a maximum of 100 and a minimum of 0 points in this questionnaire. there is a positive correlation between the score and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Volkan Deniz, Principal Investigator — Cukurova University
Locations (1):
- Volkan Deniz, Ankara, Turkey (Türkiye)